CLINICAL TRIAL: NCT02279329
Title: Longitudinal Study of 3He and 129Xe Magnetic Resonance Imaging in Chronic Obstructive Pulmonary Disease
Brief Title: Longitudinal Study of Helium-3 and Xenon-129 Magnetic Resonance Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Grace Parraga (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Dr. Grace Parraga, PhD, Scientist. Robarts Research Institute, University of Western Ontario, Canada
Organization: Western University, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ROB0018
Record Dates: First submitted 2014-10-24; First posted 2014-10-31 (Estimated); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: COPD; Bronchiectasis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD and Bronchiectasis Patients (Other): All enrolled COPD and Bronchiectasis patients will undergo Pulmonary Function Tests, Hyperpolarized Helium MRI, chest CT, 6-Minute Walk Test, and complete questionnaires at up to 8 visits over 2-3 years.
  Interventions: Other: Hyperpolarized Helium MRI

INTERVENTIONS:
Other: Hyperpolarized Helium MRI — Hyperpolarized helium-3 (3He) magnetic resonance imaging (MRI) has recently emerged as another research approach for the non-invasive measurement of lung structure and function, including conduction of gas through airways and into airspaces. Preliminary studies suggest that 3He MRI may be ideally suited for longitudinal COPD research, which is a likely target application of this novel technology. 3He MRI provides a complementary and alternative method for evaluating COPD and may be superior to CT because it allows simultaneous visualization of both airway and airspace structure and function.

SUMMARY:
Subjects male and female aged 50-85 with a clinical diagnosis of chronic obstructive pulmonary disease (COPD) or Bronchiectasis, or those with ≥ 10 pack/years smoking history will be imaged with CT and MRI for the development of tools to quantify and validate longitudinal in vivo magnetic resonance imaging phenotypes of COPD and Bronchiectasis.

DETAILED DESCRIPTION:
COPD patients will be stratified into four groups: Gold Stage 0, Gold Stage I, Gold Stage II, and Gold Stage III. During a single 2-2 ½ hour visit, patient subjects will perform some or all of: 1) spirometry pre-and-post salbutamol and plethysmography, Lung Clearance Index, Airway Oscillometry (Airwave Oscillometry measures the mechanics of the respiratory system by superimposing a gentle multi-frequency airwave onto the patient's respiratory airflow. Measurements take no longer than 16 seconds and the patient simply breathes normally into a disposable mouthpiece for the duration of the test.) 2) 6MWT (including Borg questionnaire pre-and post-walk), 3) health status evaluation using a self-administered SGRQ and MMRC (Modified Medical Research Council dyspnea scale) 4) CT, and, 5) 3He MRI.

Subjects will first provide written informed consent and then be screened for MRI compatibility and will complete: 1) Spirometry pre-salbutamol, SGRQ after inhaling 2-4 puffs (200-400μg) of the short-acting bronchodilator (eg. Salbutamol), 2) MRI, 3) CT. (Subjects will be taken by wheelchair to and from University Hospital, LHSC to decrease the potential for dynamic hyperinflation), 4) plethysmography and spirometry within 1 ½ hours of salbutamol. Vital signs will be performed. Because it is impossible to schedule imaging at the same time-point post-bronchodilator, subjects will be randomized to MR or CT 30 minutes post-salbutamol (1:1 ratio), to minimize bias.

ELIGIBILITY:
Inclusion Criteria:

* Subjects male and female aged 50-85 with either A) a clinical diagnosis of COPD or Bronchiectais or B) >10 pack/year smoking history
* Subject understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent
* Subject must be able to perform a breathhold for 16s.
* Subject is judged to be in otherwise stable health on the basis of medical history
* Subject is ambulatory and can perform the 6MWT
* Subject able to perform reproducible pulmonary function testing (i.e., the 3 best acceptable spirograms have FEV1 values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater.)
* FEV1 >25% predicted
* FVC > 25% predicted and >0.5L

Exclusion Criteria:

* Patient is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material.
* Subject has a daytime room air oxygen saturation <90% while lying supine.
* Patient is unable to perform spirometry or plethysmography maneuvers
* Patient is pregnant
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.
* Subject has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants.)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-05 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Ventilation Defect Percent (VDP) | 3 years
  VDP is a widely used noble gas MRI biomarkers that is calculated by normalizing ventilation defect volume to the thoracic cavity
Apparent Diffusion Coefficients (ADC) | 3 years
  Diffusion weighted noble gas MRI provides a way to quantify pulmonary microstructure by sensing the movements of inhaled gas atoms. The "apparent" dif fusion coefficient (ADC) during the diffusion time interval can be used to reflect the extent of alveolar restriction of gas atom movements, providing a surrogate measurement of airspace dimensions.

SECONDARY OUTCOMES:
Six Minute Walk Distance (6MWD) | 3 years
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes.
St. George's Respiratory Questionnaire (SGRQ) | 3 years
  Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.
Spirometry | 3 years
  Spirometry is a common office test used to assess how well your lungs work by measuring how much air you inhale, how much you exhale and how quickly you exhale.

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Salerno M, de Lange EE, Altes TA, Truwit JD, Brookeman JR, Mugler JP 3rd. Emphysema: hyperpolarized helium 3 diffusion MR imaging of the lungs compared with spirometric indexes--initial experience. Radiology. 2002 Jan;222(1):252-60. doi: 10.1148/radiol.2221001834. PMID 11756734
- [Background] Evans A, McCormack D, Ouriadov A, Etemad-Rezai R, Santyr G, Parraga G. Anatomical distribution of 3He apparent diffusion coefficients in severe chronic obstructive pulmonary disease. J Magn Reson Imaging. 2007 Dec;26(6):1537-47. doi: 10.1002/jmri.21205. PMID 17968961
- [Background] Mathew L, Evans A, Ouriadov A, Etemad-Rezai R, Fogel R, Santyr G, McCormack DG, Parraga G. Hyperpolarized 3He magnetic resonance imaging of chronic obstructive pulmonary disease: reproducibility at 3.0 tesla. Acad Radiol. 2008 Oct;15(10):1298-311. doi: 10.1016/j.acra.2008.04.019. PMID 18790402
- [Derived] Kooner HK, Wyszkiewicz PV, Matheson AM, McIntosh MJ, Abdelrazek M, Dhaliwal I, Nicholson JM, Kirby M, Svenningsen S, Parraga G. Chest CT Airway and Vascular Measurements in Females with COPD or Long-COVID. COPD. 2024 Dec;21(1):2394129. doi: 10.1080/15412555.2024.2394129. Epub 2024 Sep 2. PMID 39221567
- [Derived] Sharma M, Wyszkiewicz PV, Matheson AM, McCormack DG, Parraga G. Chest MRI and CT Predictors of 10-Year All-Cause Mortality in COPD. COPD. 2023 Dec;20(1):307-320. doi: 10.1080/15412555.2023.2259224. Epub 2023 Sep 22. PMID 37737132
- [Derived] Wyszkiewicz PV, Sharma M, Desaigoudar V, Cunningham IA, McCormack DG, Abdelrazek MA, Kirby M, Parraga G. Reduced Total Airway Count and Airway Wall Tapering after Three-Years in Ex-Smokers. COPD. 2023 Dec;20(1):186-196. doi: 10.1080/15412555.2023.2222831. PMID 37395048
- [Derived] Capaldi DPI, Guo F, Xing L, Parraga G. Pulmonary Ventilation Maps Generated with Free-breathing Proton MRI and a Deep Convolutional Neural Network. Radiology. 2021 Feb;298(2):427-438. doi: 10.1148/radiol.2020202861. Epub 2020 Dec 8. PMID 33289613
- [Derived] MacNeil JL, Capaldi DPI, Westcott AR, Eddy RL, Barker AL, McCormack DG, Kirby M, Parraga G. Pulmonary Imaging Phenotypes of Chronic Obstructive Pulmonary Disease Using Multiparametric Response Maps. Radiology. 2020 Apr;295(1):227-236. doi: 10.1148/radiol.2020191735. Epub 2020 Feb 25. PMID 32096708